CLINICAL TRIAL: NCT01839825
Title: Randomized Comparative Study of QuietCare (Motion Sensor System) in Elderly Subjects Living in Assisted/ Independent Living Facilities
Brief Title: Comparative Study of QuietCare
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Center for Geriatrics and Gerontology, Japan (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Takayuki Hosoi, Director, Clinical Research and Development, National Center for Geriatrics and Gerontology, Japan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 109-2012-GES-0001
Record Dates: First submitted 2013-03-30; First posted 2013-04-25 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-09

CONDITIONS: Elderly People; Living Alone in a Residence With Care Giver
Keywords: elderly; fall; acute illness; care giver

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- QuietCare (Experimental): QuieCare system installed
  Interventions: Device: QuietCare
- control (No Intervention): no system installed

INTERVENTIONS:
Device: QuietCare
  Other Names: passive monitoring system using infrared
  Arms: QuietCare

SUMMARY:
The objective of the study is to examine the efficacy and safety of QuietCare in a randomized, open study in elderly subjects living in assisted/ independent living facilities for 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. ability to move independently or by using a walker (without assistance) inside
2. residents using a single room, age 65 or older, of either sex

Exclusion Criteria:

* people who use wheel chairs,
* people who are bed-ridden

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-12; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Changes in score of Care Service Quetionnaire | The observation period is 6 months.
  * improvement in care level assessment
  * improvement in care plannning
  * improvement in communication among staff
  * improvement in communication with residents and their family
Time required for staff to respond to events | The observation period is 6 months.
Incidence of falls | The observation period is 6 months

SECONDARY OUTCOMES:
Fee for medical and nursing care treatments | The observation period is 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Home Ogori, Fukuoka, Fukuoka, Japan